CLINICAL TRIAL: NCT04001413
Title: Phase II, Adjuvant Therapy for High-Risk HPV 16-Positive Oropharynx Cancer Patients With Durvalumab (MEDI4736) and MEDI0457 (INO-3112)
Brief Title: Therapy for High-Risk HPV 16-Positive Oropharynx Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1918; IRB00179194 (Other: JHM IRB)
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma; Oropharynx Cancer; HPV-Related Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — MEDI0457; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Observational (No Intervention): No intervention, observational arm.
- Arm B: Durvalumab Alone (Experimental): Durvalumab will be administered as an IV Infusion.
  Interventions: Drug: Durvalumab
- Arm C: MEDI0457 and Durvalumab (Experimental): MEDI0457 is an injection. Durvalumab will be administered as an IV Infusion.
  Interventions: Drug: MEDI0457; Drug: Durvalumab

INTERVENTIONS:
Drug: MEDI0457 — MEDI0457 is an investigational drug that will be administered with the Cellectra Device in this study
  Other Names: INO-3112
  Arms: Arm C: MEDI0457 and Durvalumab
Drug: Durvalumab — Durvalumab is an investigational drug in this study.
  Other Names: MEDI4736
  Arms: Arm B: Durvalumab Alone; Arm C: MEDI0457 and Durvalumab

SUMMARY:
Combination immune checkpoint inhibitor and DNA vaccine will result in clearance of HPV DNA biomarkers (oral and/or plasma) for patients with persistent HPV-16 E6/E7 DNA (HPV biomarker) after treatment with curative intent.

DETAILED DESCRIPTION:
Objectives:

Primary Objectives:

To determine whether combination immune checkpoint inhibitor, alone or together with a DNA vaccine will result in clearance of HPV biomarkers for patients at risk of disease progression.

Secondary Objective(s):

1. To evaluate the time to progression among patients with detectable HPV DNA when treated with the durvalumab/MEDI0457 versus durvalumab monotherapy versus observation.
2. To assess the toxicity of durvalumab and MEDI0457 in the adjuvant setting.

Exploratory Objective(s):

1. To determine whether anti-PD-L1 alone or together with an HPV DNA vaccine will enhance HPV E6/E7-specific and/or mutation-associated neoantigen (MANA)-specific T cell responses and whether these responses correlate with enhanced clearance of HPV as measured by DNA in oral rinses and/or plasma.
2. To determine whether anti-PD-L1 alone or together with an HPV DNA vaccine will enhance HPV 16 E6/E7-specific IgG and whether these responses correlate with enhanced clearance of HPV as measured by DNA in oral rinses and/or plasma

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Men and women >or = 18 years at the time of study entry.
* Histologically or cytologically proven HPV16-positive or p16-positive oropharyngeal squamous cell carcinoma.
* Eastern Cooperative Oncology Group (ECOG) 0-1 (Appendix A)
* Completion of primary therapy curative intent )surgery based or radiation based) within the past year (date of last treatment + 1 year) OR newly diagnosed with a plan for treatment with curative intent OR currently in primary treatment with curative intent.
* Body weight or = 30kg
* Adequate organ function as follows:
* Absolute neutrophil count (ANC) > or = 1000/mm3
* Platelet count > or = 75 x 109/L(> or = 75,000 per mm3)
* Hemoglobin > or =9 g/dL
* Creatinine < or = 1.5 x institutional ULN or creatinine clearance (CrCI) > or = 40mL/min (if using Cockcroft-Gault formula below):

Female CrCI = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCI= (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL

* Total Bilirubin < or = 1.5 x institutional ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
* AST(SGOT)/ALT(SGPT) < or = 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be < or = 5x ULN
* Sexually active fertile men must use effective barrier birth control if their partners are WOCBP for up to 217 days after the last dose of durvalumab.
* The effects of Durvalumab and MEDI0475 on the developing human fetus are unknown. Women of child-bearing potential (WOCBP) and mes must agree to use at least one highly effective method of contraception (hormonal or barrier method form of birth control; abstinence) prior to study entry and for the duration of study participation and for up to 217 days after the last dose of Durvalumab or MEDI0457.
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she must inform her treating physician immediately.
* WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within two weeks of screening.
* Women must not be breastfeeding
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women > or =50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form. Voluntary signed and dated IRB/IEC guidelines must be obtained before the performance of any protocol related procedures that are not part of normal care.
* Subjects must be competent to report AEs, understand the drug dosing schedule and use of medications to control AEs.
* Individuals of all races and ethnic groups are eligible for this trial. There is no bias towards age, gender or race in the clinical trial outlined. This trial is open to accrual of men and women who meet the inclusion/exclusion criteria outlined.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during or after primary therapy.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Any unresolved toxicity NCI CTCAE Grade > or = 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in inclusion criteria.

  * Patients with Grade > or = 2 neuropathy will be evaluated on a case-by-case basis after consultation with Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Subjects with a previous diagnosis of another primary malignancy are excluded with the exception of

  * Malignancy treated with curative intent and with no known active disease > or = 3 years and of low potential risk of recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Thyroid or salivary cancer
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]. The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with study physician
  * Patients with celiac disease controlled by diet alone
  * Patients with stable, inactive rheumatoid arthritis
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of active primary immune deficiency
* Active infection including:

  * tuberculosis (clinical evaluation that includes history, physical examination and radiographic findings, and TB testing in line with local practice).
  * Hepatitis B and or hepatitis C, (positive tests for hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA) or
  * Patients with a past or resolved HBV infection (defined as the absence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
  * human immunodeficiency virus (positive HIV 1/2 antibodies).
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Active systemic infection requiring therapy.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent C. Corticosteroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not received live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
* Use of anticoagulants and irreversible platelet inhibitors (e.g. clopidogrel, prasugrel, ticagrelor, etc.) are not allowed. Low dose aspirin for cardiac prophylaxis is allowed.
* Subjects are excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Female patients who are pregnant or intend to become pregnant, breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 217 days after the last dose of durvalumab monotherapy.
* Men with female partners (WOCBP) that are not willing to use contraception from screening to 217 days after the last dose of durvalumab monotherapy.
* Unable to follow up per study schedule.
* Patient is 1 year or greater from completion of primary treatment.
* Prisoners or subjects who are involuntarily incarcerated or compulsorily detained for treatment of either psychiatric or physical (e.g. infectious disease) illness.
* Patients weighing <30kg at time of screening are to be excluded from enrollment.
* Prior therapy with an anti-PD-1, anti-PD-L1, including durvalumab anti-PDL-2, or anti-CTLA-4 antibody (or any other antibody targeting T cell co-regulatory pathways).
* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events. For example, prior symptomatic pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Number of participants in whom there is clearance of Human Papiloma Virus (HPV) biomarkers post-intervention | Up to 5 years

SECONDARY OUTCOMES:
Time to Progression | Up to 5 years
  Time until progression, followed for up to five years, among patients with detectable HPV DNA when treated with the durvalumab/MEDI0457 versus durvalumab monotherapy versus observation.
Safety of Study Drugs | Up to 30 days after the last dose of study drug
  Adverse events will be reviewed to determine the safety of durvalumab and MEDI0457 in the adjuvant setting. Observed Adverse events and toxicities will be tabulated by treatment group, type and grade. AEs and other toxicities will be graded using NCI Common Terminology Criteria for Adverse Events 5.0 (CTCAE).

OTHER OUTCOMES:
Clearance of HPV Measured by DNA in participants with HPV E6/E7-specific and MANA-specific T-cell response | Up to 5 years
  Clearance of HPV as measured by DNA in oral rinses and/or plasma (milliliters) in participants with HPV E6/E7-specific and mutation-associated neoantigen (MANA)-specific T-cell responses.
Clearance of HPV Measured by DNA in participants with HPV E6/E7-specific IgG | Up to 5 years
  Clearance of HPV as measured by DNA in oral rinses and/or plasma (milliliters) in participants with HPV E6/E7-specific IgG

CONTACTS AND LOCATIONS:
Overall Officials: Carole Fakhry, MD, MPH, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Mount Sinai School of Medicine, The Tisch Cancer Institute, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No